CLINICAL TRIAL: NCT05485948
Title: A Phase II Single-Arm Multicenter Study to Access Efficacy and Safety of P1101 in Chinese Polycythemia Vera Patients Who Are Intolerant or Resistance to Hydroxyurea
Brief Title: A Study to Access Efficacy and Safety of P1101 in Chinese PV Patients Who Are Intolerant or Resistance to HU
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A20-202
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Polycythemia Vera
Keywords: Ropeginterferon alpha-2b; Polycythemia Vera; Hydroxyurea; P1101
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with P1101 (Experimental): Subjects who meet all the inclusion criteria and do not meet any of the exclusion criteria will start treatment with P1101. The study drug will be subcutaneously injected once every 2 weeks, with the target dose being 500 µg. Subjects will receive an initial dose of 250 µg at Week 0, a medium dose of 350 µg at Week 2, a target dose of 500 µg at Week 4, and a maintenance dose of 500 µg from the subsequent week until Week 52. If the dose needs to be adjusted due to safety or tolerability consideration, it is allowed to be adjusted to the previous dose, but the target dose is preferred to be maintained during the treatment period.
  Interventions: Drug: Ropeginterferon alfa-2b

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b — Initial dose of 250 µg at Week 0, a medium dose of 350 µg at Week 2, a target dose of 500 µg at Week 4, and a maintenance dose of 500 µg until Week 52.
  Other Names: BESREMI

SUMMARY:
This study is a phase II single-arm study designed to evaluate the efficacy and safety of P1101 in Chinese PV patients who are intolerance or resistance to HU.

DETAILED DESCRIPTION:
Eligible subjects will be treated with P1101 at a starting dose of 250 µg at Week 0, a medium dose of 350 µg at Week 2, a target dose of 500 µg at Week 4, and a maintenance dose of 500 µg from the subsequent week until Week 52. At Week 24 (Month 6), the primary study endpoint, i.e., the phlebotomy- or erythrocytapheresis-free CHR rate, will be analyzed.

For subjects who switch from previous HU treatment to P1101 (for subjects who are currently receiving HU treatment), the dose should be gradually reduced during the screening period (adjusted by the investigator based on clinical practice); the HU treatment should be ended within up to 4 weeks of P1101 treatment, and HU should be prohibited after 4 weeks of P1101 treatment.

During the treatment period, subject visits are scheduled for once every 2 weeks. The end of treatment (EOT) visit will be performed at Week 52 or early termination of the study, and the end of study (EOS) visit will be performed at 28 days after the EOT visit.

Data analyses will be performed after all subjects complete 24 weeks of treatment, and a clinical trial report written, and the new drug application is submitted accordingly. An end-of-study statistical analysis will be performed after all the subjects have completed all visits as per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years at the time of signing the informed consent form;
* Patients diagnosed with PV according to the 2016 World Health Organization (WHO) criteria;
* According to the 2020 Guidelines of Chinese Society of Clinical Oncology (CSCO) on Diagnosis and Treatment of Hematological Malignancies, PV patients who are HU resistant or intolerant must meet at least one of the following criteria;

  1. Drug resistance: 3 months of treatment at HU doses above 2 g/d

     1. Phlebotomy is still required to maintain Hct <45%;
     2. Failure to control the bone marrow proliferation (such as platelet count >400x10^9/L and white blood cell count >10x10^9/L);
     3. spleen shrinkage of less than >50%;
  2. Intolerance

     1. At the minimum dose of HU required to achieve complete or partial clinical hematologic response, the absolute neutrophil count (ANC) <1x10^9/L or PLT <100x10^9/L or HGB <100 g/L;
     2. At any dose of HU treatment, the patient develops lower limb ulcers or other intolerable non-hematologic toxicity, such as skin mucosal manifestations (dark skin, teeth or nails; oral ulcers, mucositis; skin ulcers, rash, and other symptoms), gastrointestinal complaints (nausea, loss of appetite, indigestion, vomiting, abdominal pain, constipation, and other symptoms), pneumonia, fever, etc.
* Have not received interferon therapy previously; or have negative anti-P1101 binding antibody at screening, and the washout time between the last dose of interferon and the first dose of the study drug should not be shorter than 14 days;
* With good liver function at screening, which is defined as total bilirubin ≤1.5 × upper limit of normal (ULN), international normalized ratio (INR) ≤1.5 × ULN, albumin >3.5 g/dL, alanine aminotransferase (ALT) ≤2.0 × ULN, and aspartate aminotransferase (AST) ≤2.0 × ULN;
* Hemoglobin (HGB) ≥10 g/dL for females, and hemoglobin (HGB) ≥11 g/dL for males at screening;
* Neutrophil count ≥1.5x10^9/L at screening;
* Creatinine clearance rate ≥40 mL/min at screening (according to the Cockcroft-Gault formula);
* Males and females of childbearing potential, as well as all the females with a menopause duration of less than 2 years, must consent to use acceptable contraceptive methods within 28 days after the last dose of the study drug;
* The patient or the patient's guardian signs the written informed consent, and the patient is able to comply with the study requirements.

Exclusion Criteria:

* Patients with symptomatic splenomegaly;
* Any contraindications to interferon α or hypersensitivity to interferon α;
* With severe or serious diseases that the investigator determines may affect the patient's participation in this study;
* History of major organ transplantation;
* Pregnant or breastfeeding women;
* Patients with any other diseases that the investigator determines will affect the study results or may weaken the compliance to protocol, including but not limited to:

  1. Prior or current autoimmune thyroid disease, but patients with oral thyroxine replacement therapy could be enrolled;
  2. Other documented autoimmune diseases (such as hepatitis, immune thrombocytopenia [ITP], scleroderma, psoriasis or any autoimmune arthritis);
  3. Clinically significant pulmonary infiltration, infectious pneumonia and non-infectious pneumonia, or a past history of interstitial pneumonia at screening;
  4. Active infection with systemic manifestations (e.g., presence of bacteria, fungi and human immunodeficiency virus [HIV], excluding hepatitis B [HBV] and/or hepatitis C [HCV] at screening);
  5. With evidence of severe retinopathy (e.g., cytomegalovirus [CMV]-induced retinitis, macular degeneration) or clinically significant eye diseases (due to diabetes or hypertension);
  6. With clinically significant depression or a history of depression;
  7. Previously had suicidal attempts or has any risk for suicidal tendency at screening.
* Poorly controlled diabetes;
* Thromboembolic complications caused by PV and active abdomina hemorrhage;
* History of any malignancy tumors (except stage 0 chronic lymphocytic leukemia [CLL], cured basal cell carcinoma, squamous cell carcinoma and superficial melanoma) in the past 5 years;
* History of alcohol or drug abuse in the past year;
* History or evidence of post polycythemia vera-myelofibrosis (PPV-MF), essential thrombocythemia, or any non-PV MPN;
* Presence of blast cells in the peripheral blood in the past 3 months;
* Use any investigational drugs or investigational drug combinations within 4 weeks before the first dose of the study drug, or have not yet recovered from the effects caused by any previously administered investigational drug.

Unless with contraindications, acetylsalicylic acid will be considered as background treatment of this study. The following are contraindications to low-dose acetylsalicylic acid: history of allergies to Bayaspirin or any preparations of salicylic acid, peptic ulcer, bleeding tendency, aspirin-induced asthma (asthma attack caused by non-steroidal anti-inflammatory drugs, etc.) and its history. If any contraindications are found, other prophylactic anti-thrombotic drugs can be used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The phlebotomy- or erythrocytapheresis-free CHR rate based on the central laboratory test results evaluation | Week 24
  1. Hct <45% without the use of phlebotomy or erythrocytapheresis (without the use of phlebotomy or erythrocytapheresis within the previous 3 months);
  2. PLT count≤400x10^9/L;
  3. WBC count <10x10^9/L.

SECONDARY OUTCOMES:
The phlebotomy- or erythrocytapheresis-free CHR rate based on the evaluation of central laboratory test results | Weeks 12, 36 and 52
  1. Hct <45% without the use of phlebotomy or erythrocytapheresis (without the use of phlebotomy or erythrocytapheresis within the previous 3 months);
  2. PLT count≤400x10^9/L;
  3. WBC count <10x10^9/L.

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing Zhang, Study Director — PharmaEssentia
Locations (14):
- China (14):
  - Peking Union Medical College Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - The First Affiliated Hospital of Chongqing Medical Universit, Chongqing
  - Nanfang Hospital affiliated to Southern Medical University, Guangzhou
  - Anhui Provincial Hospital, Hefei
  - Huashan Hospital affiliated to Fudan University, Shanghai
  - Ruijin Hospital affiliated to Shanghai Jiaotong University, Shanghai
  - Shenzhen Second People's Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Institute of Hematology &Blood Diseases Hospital ,Chinese Academy of medical science & Peking Union Medical College, Tianjin
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Zhongnan Hospital affiliated to Wuhan University, Wuhan
  - The First Affiliated Hospital Zhejiang University of Medicine, Zhejiang
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin J, Zhang L, Qin A, Wu D, Shao Z, Bai J, Chen S, Duan M, Zhou H, Xu N, Zhang S, Zuo X, Du X, Wang L, Li P, Zhang X, Li Y, Zhang J, Wang W, Shen W, Zagrijtschuk O, Urbanski R, Sato T, Xiao Z. A new dosing regimen of ropeginterferon alfa-2b is highly effective and tolerable: findings from a phase 2 study in Chinese patients with polycythemia vera. Exp Hematol Oncol. 2023 Jun 21;12(1):55. doi: 10.1186/s40164-023-00415-0. PMID 37344895
- [Derived] Jin J, Qin A, Zhang L, Shen W, Wang W, Zhang J, Li Y, Wu D, Xiao Z. A phase II trial to assess the efficacy and safety of ropeginterferon alpha-2b in Chinese patients with polycythemia vera. Future Oncol. 2023 Apr;19(11):753-761. doi: 10.2217/fon-2022-1141. Epub 2023 May 2. PMID 37129584